CLINICAL TRIAL: NCT02136602
Title: Interventricular Cardiac Septal Thickness in Fetus of Diabetic Mother Correlated to Postnatal Outcome
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, heba elsyed, helsayed, Ain Shams University
Other Study IDs: hct 4321
Record Dates: First submitted 2013-11-06; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Maternal Diabetes Mellites Effect on Fetus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: None Retained — pregnant over 35 weeks. medically free.single intrauterine pregnancy
Oversight: Data Monitoring Committee: No

SUMMARY:
Good glycemic control is superior to poor glycemic control in reducing risk of interventricular septal thickness among fetuses of diabetic mothers.

DETAILED DESCRIPTION:
Thick Interventricular septum is thought to be related to poor glycemic control during pregnancy, and it causes variable degree of left ventricular outflow obstruction and hypertrophic cardiomyopathy.

Hypertrophic cardiomyopathy requires specific management as digoxin and inotropic agents usually used in heart failure are contraindicated.

So high index of suspicion is required in fetus of diabetic mother having thick Inter ventricular septum.

ELIGIBILITY:
Inclusion Criteria:

* above 35 weeks pregnancy
* diabetic mothers
* single intrauterine pregnancy

Exclusion Criteria:

* any other medical disorder

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women with diabetes mellites
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To study interventricular septal thickness in fetus of diabetic mother and correlate it with good glycemic control. | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed M Elsafty, obs&gyn lecturer., Study Director — Ain Shames university
Locations (1):
- AinShamsU, Cairo, Egypt